CLINICAL TRIAL: NCT06004648
Title: Comparison of Anesthetic and Analgesic Efficacy of Selective Trunk and Supraclavicular Brachial Plexus Blocks in Upper Extremity Surgery
Brief Title: Comparison of Selective Trunk and Supraclavicular Brachial Plexus Blocks
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Döndü Genc Moralar, head of anesthesiology,Clinical Professor, Gaziosmanpasa Research and Education Hospital
Other Study IDs: 107
Record Dates: First submitted 2023-08-14; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Upper Extremity Problem
Keywords: nerve block; Pain, Postoperative; Anesthetics, Local
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Supraclavicular nerve block: The high- frequency linear USG probe will be placed in the supraclavicular fossa pointing caudally, and the subclavian artery will be localized by moving it medially and laterally. A characteristic honeycomb plexus will be visualized in the lateral and superficial subclavian artery. Vascular structures will be detected using color Doppler, the first rib will be visualized as hyperechoic structure. After the pleura, which makes a
  sliding movement through the patient's breathing is detected, a 22 gauge, 80 mm scale peripheral block needle will be directed from the lateral to the medial by an in-plane technique. After the sheath punctured, nerves will be determined with triceps, biceps, and wrist motor activity by using a nerve stimulator, and then 15 ml of 0.5% bupivacaine will be injected between the 1st rib and the lower trunk.
  Interventions: Procedure: Upper extremity surgery
- Selective Trunk Block: Sequential ultrasound imaging technique (SUIT) will be used which is shown successfully in identifying individual elements of the brachial plexus. The neural complex of the upper trunk, middle trunk, and C8 ventral ramus, which are superficial to the T1 TP-1.rip complex will be defined. The first injections contains 8 ml and 7 ml 0.5% bupivacaine will be made as, close to the upper trunk(8ml) and middle trunk(7ml) in the interscalene groove. Then the needle will be completely withdrawn.The ultrasound probe will be placed caudally in the supraclavicular fossa. After providing the optimal view of the lower trunk in the corner pocket, 10 ml of 0.5% bupivacaine will be injected between the first rib and lower trunk.
  Interventions: Procedure: Upper extremity surgery

INTERVENTIONS:
Procedure: Upper extremity surgery — Comparison of 2 different peripheral nerve blocks

SUMMARY:
There are different methods in brachial plexus blocks for hand, wrist, forearm, and elbow operations. In this study, the anesthetic efficacy of the ultrasound-guided selective truncus methods and the supraclavicular methods for brachial plexus blocks in upper extremity surgeries will be compared.

DETAILED DESCRIPTION:
Currently, brachial plexus block performed with various approaches is preferred to general anesthesia due to its advantages in upper extremity surgeries. These advantages can be listed as protecting the patient's consciousness, minimum effect on breathing, reducing airway interventions, enabling long-term postoperative pain control, reducing opioid-related side effects, limiting metabolic and endocrine changes due to surgery, and early discharge of hospital. The supraclavicular approach has a rapid onset of block and a high success rate. Close proximity to the pleura is the main disadvantage, but the widespread use of USG in peripheral blocks has also reduced the risk of complications related to this proximity. In the selective truncus approach defined by Manoj Kumar Karmakar in 2020, three trunks of the brachial plexus can be identified separately and selectively blocked under ultrasound guidance. It has been suggested that sensory/motor block occurs in all ipsilateral upper extremity dermatomes except T2 by selective blocking of the upper, middle, and lower trunks. In this study, the selective trunk method and the supraclavicular method will be compared.

Patients who will undergo upper extremity elbow and below-elbow surgery in the orthopedics and traumatology operating room will be included in the study. The primary aim of the study is to compare the success rates of supraclavicular and selective truncus blocks in patients scheduled for hand, wrist, forearm, and elbow surgery. Comparisons will be made by measuring the first analgesic time after surgery. Secondary aims are sensory and motor block success rates between the two methods. The block application time, preparation time for surgery, number of needle insertions, tourniquet pain, diaphragmatic paralysis rate, complications (vascular puncture, paresthesia, horner's syndrome, hoarseness, local anesthetic toxicity, pneumothorax) patient satisfaction, surgeon satisfaction and total analgesic amount at the end of the postoperative 12 and 24 hours will be recorded.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing upper extremity elbow and below-elbow surgery in the orthopedics and traumatology operating room

Exclusion Criteria:

* Patient's refusal
* ASA IV,
* Pregnancy,
* Neuromuscular disease,
* Peripheral neuropathy
* Bleeding disorders,
* Local anesthetic allergy,
* Infection in the block area
* Operations without using a tourniquet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthopedic surgery patients between 18-65 years of age who needs upper extremity elbow and below-elbow surgery
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
peripheral block success | T1: 12 hours after surgery, T2: 24 hours after surgery
  primary aim of the study is to compare the success rates of supraclavicular and selective truncus blocks in patients scheduled for hand, wrist, forearm, and elbow surgery. Comparison will be made by measuring the first analgesic time after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: ZÜHAL ÇAVUŞ, Study Chair — gaziosmanpasa TREH
Locations (1):
- Zühal Çavuş, Istanbul, Gaziosmanpaşa, Turkey (Türkiye)